CLINICAL TRIAL: NCT01884207
Title: Multiparametric Characterization of Orbital Tumors by MRI
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sa-Ra Ro, doctoral candidate, Charite University, Berlin, Germany
Other Study IDs: MCOT_03_05
Record Dates: First submitted 2013-06-06; First posted 2013-06-21 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Orbital Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- orbital tumors
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI

SUMMARY:
Prospective study on patients with orbital tumors of unknown origin. Aim of the study is to differentiate benign from malignant tumors upon MR imaging. Magnetic resonance imaging of the orbit will be performed including standard morphological sequences and advanced sequence techniques. These advanced sequence techniques may allow to differentiate benign from malignant tumors based on their cellularity and vascularity (diffusion and perfusion imaging). These MRI data will be analysed and the level of diffusion and perfusion will be measured and compared to the histological findings. Cut-off values of diffusion and perfusion will be calculated that allow to separate benign from malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* non-diagnosed orbital tumors

Exclusion Criteria:

* any metal implants, non-MRI compatible
* age below 18
* pregnancy
* recent surgery
* recent severe medical diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with orbital tumors
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
multiparametric characterization of orbital tumors by MRI | 24 months
  The level of diffusion and perfusion (multiparametric characterization) of the orbital tumors will be measured and the outcome measure is the ability of diffusion and perfusion imaging to predict malignancy. These parameters will be compared to histopathology in terms of separating benign vs. malignant tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany